CLINICAL TRIAL: NCT01530945
Title: Mapping Multidimensional Illness Trajectories of Patients With ESKD
Brief Title: Mapping Multidimensional Illness Trajectories of Patients With End-stage Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01NR013359 (NIH); R01NR013359 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients with end-stage kidney disease (ESKD) must manage not only the demands of dialysis and comorbid conditions but also associated symptoms and acute life-threatening events that contribute to functional limitations and increased risk of mortality. Yet little is known about the trajectories of quality of life dimensions in patients with ESKD when they experience acute life-threatening episodes, to guide palliative care for this population. In this prospective, descriptive study, we will identify trajectories of symptoms, physical functioning, psychosocial needs, and emotional and spiritual well-being in 200 patients with ESKD who are at a high risk of experiencing acute life-threatening events and mortality within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older;
* receiving either Hemodialysis or Peritoneal dialysis
* on dialysis either < 3 months or ≥ 6 months with a Charlson Comorbidity Index (CCI) score ≥ 5

Exclusion Criteria:

* Patients who are enrolled in hospice or too sick to participate in questionnaire completion will not be eligible.
* Kidney transplant candidates will be excluded because their illness trajectories after transplant are likely to differ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESKD patients who have been on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Symptoms, physical functioning, psychosocial needs, spiritual well-being, cognitive functioning | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, PhD, RN, FAAN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals and outpatient dialysis clinics, Chapel Hill, North Carolina, United States